CLINICAL TRIAL: NCT06919016
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of the V3-region Directed Immunogens DV700P-RNA (Prime) Followed by DV701B1.1-RNA (Boost) in Adult Participants Without HIV
Brief Title: A Study to Evaluate the Safety and Immunogenicity of the V3-region Directed Immunogens DV700P-RNA Followed by DV701B1.1-RNA in Adults Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 321
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): DV700P-RNA: 50 mcg at weeks 0, 8, and 24 DV701B1.1-RNA: 50 mcg at week 40
  Interventions: Biological: DV700P-RNA; Biological: DV701B1.1-RNA
- Group 2 (Experimental): DV700P-RNA: 100 mcg at weeks 0, 8, and 24 DV701B1.1-RNA: 100 mcg at week 40
  Interventions: Biological: DV700P-RNA; Biological: DV701B1.1-RNA
- Group 3 (Experimental): DV700P-RNA: 150 mcg at weeks 0, 8, and 24 DV701B1.1-RNA: 150 mcg at week 40
  Interventions: Biological: DV700P-RNA; Biological: DV701B1.1-RNA

INTERVENTIONS:
Biological: DV700P-RNA — Intramuscular (IM) injection
Biological: DV701B1.1-RNA — IM injection

SUMMARY:
This is a phase 1, first-in-human (FIH) trial for two vaccines, DV700P-RNA and DV701B1.1-RNA. This means it is the first time these study products are being tested in people.

The purpose of this study is to see if the study products are safe, if people are able to take them without becoming too uncomfortable, and how a person's immune system responds to them (a person's immune system protects them from infections and disease).

Forty-five volunteers without HIV and in overall good health, aged 18 to 55 years, will be enrolled and be in this study for about 16 months (about 12 visits), Study procedures will include blood draws, injections, and the collection of white blood cells and cells from their lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Understands the study and agrees to complete the consent process.
* Can attend all clinic visits until the end of the study.
* Agrees to follow all study procedures.
* Will not join another study with experimental treatments during this trial, unless approved by both study sponsors.
* Generally healthy according to the study doctor.
* Physical exam and lab results show no major issues that could affect safety or study results.
* Agrees to discuss HIV risk and prevention.
* Hemoglobin levels: at least 11.0 g/dL for women and 13.0 g/dL for men.
* White blood cell count between 2,500 to 12,000/mm³ (higher levels okay if health is otherwise good and approved).
* Platelet count between 125,000 to 550,000/mm³.
* ALT enzyme level less than 2.5 times the upper limit of normal.
* Serum creatinine level within 1.1 times the upper limit of normal.
* Serum calcium level at least 8.5 mg/dL.
* Blood pressure within acceptable range (systolic 90-140 mmHg, diastolic 50-90 mmHg), with average below 140/90 mmHg and no single reading over 160/100 mmHg.
* Negative HIV test.
* Negative for Hepatitis C.
* Negative for Hepatitis B.
* Women who can become pregnant must use effective contraception from 21 days before joining the study until 8 weeks after the last vaccination and must have a negative pregnancy test on enrollment day.
* Women of pregnancy potential must agree not to seek pregnancy through methods like IVF from 21 days before joining the study until 8 weeks after the last vaccination.

Exclusion Criteria:

* Breastfeeding or pregnant.
* Body mass index (BMI) of 40 or higher, unless in good health and approved.
* Diabetes, unless it is well-controlled Type 2 diabetes or gestational diabetes.
* Previous or current investigational HIV vaccine recipients (placebo recipients are allowed).
* Received non-HIV investigational vaccines within the last year, unless they are now licensed or authorized.
* Immunodeficiency or medications that impair immune response, such as high-dose steroids.
* Received blood products or immunoglobulin within 16 weeks before enrollment.
* Received certain vaccines within the last 4 weeks before enrollment.
* Received other vaccines within 14 days before enrollment.
* History of myocarditis or pericarditis.
* Started allergy immunotherapy in the past year (unless stable and approved).
* Taken investigational research agents recently.
* Serious allergic reactions to any mRNA vaccine or drugs containing polyethylene glycol.
* History of hereditary or acquired angioedema.
* Any episode of hives (urticaria) within the past year.
* Chronic hives (urticaria).
* Hives previously caused by immunization.
* Bleeding disorder that would make study procedures unsafe.
* Seizures or use of seizure medications in the past 3 years.
* Absence of spleen or non-functional spleen.
* Active duty and reserve US military personnel.
* Any other significant condition that could affect safety or participation, including substance use, psychiatric disorders, recent suicide attempts, or cancer with potential for recurrence.
* Asthma that requires frequent or high-dose medication, recent emergency care, or multiple daily medications.
* History of certain immune-mediated conditions (mild, localized conditions may be okay).
* Allergy to local anesthetics like Novocaine or Lidocaine.
* Difficulty with venous access, such as history of intravenous drug use or problems with blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of local reactogenicity signs and symptoms | At days 15, 71, 183 and 295 (14 days following receipt of any study vaccine)
Incidence of systemic reactogenicity signs and symptoms | At days 15, 71, 183 and 295 (14 days following receipt of any study vaccine)
Number of participants experiencing Serious adverse events (SAEs) | Baseline through Month 22
Number of participants experiencing medically attended adverse events (MAAEs) | Baseline through Month 22
Number of participants experiencing adverse events of special interest (AESIs) | Baseline through Month 22
Number of participants experiencing adverse events (AEs) leading to early participant withdrawal or permanent discontinuation will be collected throughout the study | Baseline through Month 22
Response rate of V3G-specific IgG+ B cells, as assessed by flow cytometry | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Response rate of differential serum antibody neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses as measured by the TZM-bl assay | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Magnitude of differential serum antibody neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses as measured by the TZM-bl assay | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)

SECONDARY OUTCOMES:
Response rate of serum IgG binding antibodies to autologous and heterologous HIV Env stabilized trimers, as assessed by binding antibody multiplex assay (BAMA) | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Magnitude of serum IgG binding antibodies to autologous and heterologous HIV Env stabilized trimers, as assessed by BAMA | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Response rate of serum antibody (Ab) neutralization of heterologous tier 2 HIV-1 strains, as measured by TZM-bl assay | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Magnitude of serum Ab neutralization of heterologous tier 2 HIV-1 strains, as measured by TZM-bl assay | At weeks 26 and 42 (2 weeks after the third and fourth vaccinations)
Frequency of V3G bnAb lineage sequences, as measured by B-cell receptor (BCR) single-cell sequencing of V3G-specific IgG+ B cells | Baseline though Month 22
Epitope-specific response rates, as measured by electron microscopy-based polyclonal epitope mapping (EMPEM) | At week 42 (2 weeks after the fourth vaccinations)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Alabama Medical Center (Site ID: 31788), Birmingham, Alabama
  - The Hope Clinic of the Emory Vaccine Center CRS (Site ID: 31440), Decatur, Georgia
  - Brigham and Women's Hospital (Site ID: 30007), Boston, Massachusetts
  - Columbia P&S CRS (Site ID: 30329), New York, New York
  - University of Rochester Medical Center (Site ID: 31467), Rochester, New York
  - University of Pittsburgh (Site ID: 1001), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center (Site ID: 30352), Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS (Site ID: 30331), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No